CLINICAL TRIAL: NCT06427395
Title: A Multicenter, Open-Label, Extension Clinical Trial to Evaluate Safety and Efficacy of Saroglitazar Magnesium in Participants With Primary Biliary Cholangitis (PBC)
Brief Title: Open-Label Extension Study of Saroglitazar Magnesium in Participants With Primary Biliary Cholangitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARO.23.002
Record Dates: First submitted 2024-05-09; First posted 2024-05-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-05

CONDITIONS: Primary Biliary Cholangitis
Keywords: Saroglitazar Magnesium; Primary Biliary Cholangitis; PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — saroglitazar

STUDY DESIGN:
Intervention Model Description: Multicenter, Open-Label, phase III, safety and efficacy study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Saroglitazar Magnesium 1 mg (Experimental): Saroglitazar Magnesium 1 mg tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment (24 months).
  Interventions: Drug: Saroglitazar Magnesium 1 mg

INTERVENTIONS:
Drug: Saroglitazar Magnesium 1 mg — Saroglitazar Magnesium 1 mg will be assigned to all participants enrolled in the open label extension program

SUMMARY:
Open-Label Extension Study of Saroglitazar Magnesium in Participants With Primary Biliary Cholangitis

DETAILED DESCRIPTION:
A Multicenter, Open-Label, Extension Clinical trial to evaluate Safety and Efficacy of Saroglitazar Magnesium in Participants with Primary Biliary Cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent and agree to comply with the trial protocol
2. Participated and completed SARO.21.001, the double-blind treatment phase study

Exclusion Criteria:

1. Consumption of 2 standard drinks per day if male and 1 standard drink per day if female for 3 consecutive months (12 consecutive weeks) throughout double-blind phase till screening.
2. Participants with MELD 3.0 score of 15 or greater
3. History or presence of other concomitant liver diseases at screening:

   1. Chronic hepatitis B or C virus (HBV, HCV) infection
   2. Primary sclerosing cholangitis (PSC)
   3. Alcoholic liver disease
   4. Autoimmune hepatitis (AIH)-PBC overlap syndrome
   5. Hemochromatosis
   6. Non-alcoholic steatohepatitis (NASH) on historical biopsy
4. Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, uncontrolled ascites, encephalopathy, history of variceal bleeding or history of hepatorenal syndrome at screening.
5. Use of Thiazolidinediones or Fibrates (within 12 weeks prior to screening)
6. Use of other PPAR agonists (i.e., Elafibranor, Seladelpar), Obeticholic acid (OCA), methotrexate, budesonide and other systemic corticosteroids (Prednisone dose more than 10 mg); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid, or nitrofurantoin) (within 12 weeks prior to screening)
7. History of bowel surgery (gastrointestinal [bariatric] surgery in the preceding 1 year or undergoing evaluation for gastrointestinal surgery (bariatric surgery for obesity, extensive small-bowel resection) or orthotopic liver transplant (OLT) or listed for OLT
8. Unstable cardiovascular disease, including:

   1. Unstable angina, (i.e., new or worsening symptoms of coronary heart disease in the 12 weeks before screening and throughout the screening period), acute coronary syndrome in the 24 weeks before screening and throughout the screening period, acute myocardial infarction in the 12 weeks before screening and throughout the screening period or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, in the 24 weeks before screening and throughout the screening period
   2. History/current unstable cardiac dysrhythmias
   3. Uncontrolled hypertension at screening
   4. Stroke or transient ischemic attack in the 24 weeks before screening
9. History of intracranial hemorrhage, arteriovenous malformation, bleeding disorder, and coagulation disorders
10. An uncontrolled thyroid disorder

    1. Uncontrolled hyperthyroidism: defined as any history of hyperthyroidism that has either not been treated with either radioactive iodine and/or surgery or that has been treated with radioactive iodine and/or surgery, but has required ongoing continuous or intermittent use of thyroid hormone synthesis inhibitors (i.e., methimazole or propylthiouracil) in the 24 weeks before screening
    2. Uncontrolled hypothyroidism: defined as initiation of thyroid hormone replacement therapy or dose adjustment of replacement therapy in the 12 weeks before screening
11. History of myopathies or evidence of active muscle disease demonstrated by CPK ≥ 5 × ULN at screening
12. Any of the following laboratory values:

    1. Total bilirubin > 3 x ULN
    2. Platelets < 50 × 103/mL
    3. Albumin < 2.8 g/dL
    4. eGFR < 45 mL/min/1.73 m2
    5. ALT or AST > 250 U/L
    6. ALP > 10 × ULN
13. Participation in another interventional clinical study and receipt of any other investigational medication or medical device within 30 days or within 5 half-lives, whatever is longer, prior to screening
14. History of malignancy in the past 5 years and/or active neoplasm which may diminish life expectancy (except resolved superficial non-melanoma skin cancer, carcinomas in situ or other stable, relatively benign conditions if appropriately treated prior to screening)
15. Known allergy, sensitivity or intolerance to the study medication or formulation ingredients
16. Pregnancy-related exclusions, including:

    1. Pregnant/lactating female (including positive pregnancy test at screening)
    2. Participants agree to avoid pregnancy either by true abstinence or the use of an acceptable effective contraceptive measures for the duration of the study and for at least 1 month after the end of the study medication. Refer Appendix 9 Contraceptive Guidance.
17. History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, HIV, coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption)
18. Cirrhosis with Child-Pugh-Turcotte (CPT) class B or C having score of 7 or above at screening (Refer Appendix 11

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2027-07-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From baseline to 24 Months/EOT

SECONDARY OUTCOMES:
Proportion of participants achieving biochemical response based on the composite endpoints of ALP and total bilirubin | From baseline to Months 12 and 24/EOT
  ALP < 1.67 x ULN, ≥ 15% decrease in ALP, and total bilirubin ≤ ULN or direct bilirubin ≤ ULN relative to baseline in participants with known Gilbert's syndrome
Proportion of participants with biochemical response based on the composite endpoints of ALP and total bilirubin | From baseline to Months 12 and 24/EOT
  complete normalization of ALP. Change and percent change from baseline in ALP
Time to occurrence of the clinical outcome events in study participants with PBC | From baseline to 24 Months/EOT
  Defined as new onset or recurrence of any of the following:
  * Hospitalization for new onset or recurrence of variceal bleed
  * Hepatic encephalopathy (as defined by a West Haven score ≥2)
  * New onset ascites requiring treatment
  * Refractory ascites (requiring large volume paracentesis)
  * Spontaneous bacterial peritonitis (confirmed by culture from diagnostic paracentesis)
Time to occurrence of the clinical outcome events based on Model for End Stage Liver Disease 3.0 score | From baseline to 24 Months/EOT
  Time from enrolment to the first occurrence of Model for End Stage Liver Disease 3.0 score ≥ 15 and 25% increase from baseline as measured on 2 consecutive occasions performed at least two weeks apart with no competing etiologies identified
Time to first occurrence of Liver transplant or placement on a liver transplant list | From baseline to 24 Months/EOT
Time to the occurrence of Death | From baseline to 24 Months/EOT
  Death (liver and non-liver related)
Effect on liver enzyme parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in ALT
Effect on liver enzyme parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in AST
Effect on liver enzyme parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in GGT
Effect on liver enzyme parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in total bilirubin
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in TG
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in LDL-C
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in HDL-C
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in VLDL-C
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in total cholesterol
Effect on lipid parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in non-HDL-C
Effect on liver enzyme parameters | From baseline to Months 12 and 24/EOT
  Change from baseline in serum bile acids
Effect on disease-related symptoms | From baseline to Months 12 and 24/EOT
  Change from baseline in quality of life (Primary Biliary Cholangitis- 40) questionnaire domains Scale as Never, Rarely, Sometimes, Most of the time, and Always
Effect on disease-related symptoms | From baseline to Months 12 and 24/EOT
  Change from baseline in 5-D itch scale Score ranging from 5 to 25, where higher score represents worst itching
Effect on disease-related symptoms | From baseline to Months 12 and 24/EOT
  Change from baseline in Worst Itch NRS (numerical rating scale) scores 0-10, where 0 is no itch and 10 is worst itch imaginable
Effect on liver stiffness measurement (LSM) assessed by Liver elastography/FibroScan | From baseline to Months 12 and 24/EOT
  Change from baseline in LSM assessed by Liver elastography/FibroScan

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, Study Director — Zydus Therapeutics Inc.
Locations (28):
- United States (17):
  - Zydus US013, Los Angeles, California
  - Zydus US011, Pasadena, California
  - Zydus US043, Sacramento, California
  - Zydus US022, Aurora, Colorado
  - Zydus US037, New Haven, Connecticut
  - Zydus US027, Jacksonville, Florida
  - Zydus US006, Lakewood Rch, Florida
  - Zydus US005, Miami, Florida
  - Zydus US020, Marietta, Georgia
  - Zydus US001, Indianapolis, Indiana
  - Zydus US035, Rochester, New York
  - Zydus US002, Charlotte, North Carolina
  - Zydus US042, Houston, Texas
  - Zydus US031, Murray, Utah
  - Zydus US016, Charlottesville, Virginia
  - Zydus US039, Richmond, Virginia
  - Zydus US033, Seattle, Washington
- Argentina (6):
  - Zydus AR001, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Zydus AR007, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Zydus AR006, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Zydus AR005, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Zydus AR003, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Zydus AR004, Pilar, Buenos Aires
- Turkey (Türkiye) (5):
  - Zydus TR016, Altındağ
  - Zydus TR004, Ankara
  - Zydus TR005, Bursa
  - Zydus TR017, Cebeli
  - Zydus TR015, Melikgazi